CLINICAL TRIAL: NCT02324257
Title: An Open-Label, Multicenter, Dose-Escalation Phase I Study to Evaluate the Safety, Pharmacokinetics, and Therapeutic Activity of RO6958688, A Novel T-cell Bispecific Antibody That Targets the Human Carcinoembryonic Antigen (CEA) on Tumor Cells and CD3 on T Cells, Administered Intravenously in Patients With Locally Advanced and/or Metastatic CEA(+) Solid Tumors
Brief Title: A Study of RO6958688 in Participants With Locally Advanced and/or Metastatic Carcinoembryonic Antigen Positive Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP29541; 2014-003075-30 (EudraCT Number); RG7802 (Other: Roche)
Record Dates: First submitted 2014-12-12; First posted 2014-12-24 (Estimated); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Solid Tumors
MeSH Terms: interventions — obinutuzumab; tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I: RO6958688 (Experimental): Participants will receive single dose of RO6958688 starting from a dose of 0.05, 0.15, 0.45, 1.3, and 2.5 mg in Part I of the study.
  Interventions: Drug: RO6958688; Drug: Tocilizumab
- Part II: RO6958688 With/Without Obinutuzumab Pretreatment (Experimental): Participants will receive RO6958688 with or without obinutuzumab pretreatment QW, Q3W, or according to a combined QW/Q3W step up dosing schedule. Doses will start at 40mg and increase with each administration up to the MTD or 1200mg, whichever is lower.
  Interventions: Drug: RO6958688; Drug: Obinutuzumab; Drug: Tocilizumab

INTERVENTIONS:
Drug: RO6958688 — RO6958688 is given as an intravenous (IV) infusion as a single administration in Part I, and QW, Q3W, or as a combined QW/Q3W step up dosing regimen (cycle = 7 days in the QW regimen and cycle = 21 days in the Q3W regimen) in Part II of the study.
Drug: Obinutuzumab — Obinutuzumab is given as an IV infusion at a dose level of 2000 mg on Day -13 or 1000 mg on Days -13 and -12 prior to the treatment start with RO6958688 on Cycle 1 Day 1.
  Arms: Part II: RO6958688 With/Without Obinutuzumab Pretreatment
Drug: Tocilizumab — Tocilizumab will be administered as an IV infusion as necessary to treat adverse events.

SUMMARY:
Study BP29541 is a first-in-human, open-label, multi-center, dose-escalation Phase I clinical study of single-agent RO6958688 in participants with locally advanced and/or metastatic carcinoembryonic antigen (CEA) positive solid tumors who have progressed on standard treatment, are intolerant to standard of care (SOC), and/or are non-amenable to SOC. The study will be conducted in two parts. Part I of the study will investigate the safety and pharmacokinetics of a single dose of RO6958688 in single participant cohorts with dosing starting from a minimal anticipated biological effect level dose of 0.05 milligrams (mg) and up to a maximum dose of 2.5 mg. Part II will establish the appropriate therapeutic dose based on safety, pharmacokinetics, and the maximum tolerated dose (MTD) of RO6958688 for the once per week (QW) regimen, every three weeks (Q3W) regimen, and for the step up dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

* For dose escalation, locally advanced and/or metastatic gastrointestinal (GI) solid tumor in participants who have progressed on a standard therapy, are intolerant to SOC, and/or are non-amenable to SOC and other solid tumors expressing CEA. Only locally advanced and/or metastatic colorectal cancer participants should be included in the scheduled comparison expansion
* Radiologically measurable disease according to RECIST v1.1
* Life expectancy, in the opinion of the investigator of greater than or equal (>/=) to 12 weeks and LDH= 2.5 x ULN
* Eastern Cooperative Oncology Group Performance Status of 0-1
* All acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure must have resolved to Grade less than or equal to 1 or returned to baseline except alopecia (any grade) and Grade 2 peripheral neuropathy
* Adequate hematological, liver, and renal function
* Participants must agree to remain abstinent or be willing to use effective methods of contraception as defined in the protocol
* Non-GI solid tumors (like non-small cell lung cancer or breast cancer) should have confirmed CEA expression in tumor tissue >/= 20% of tumor cells staining with at least moderate to high intensity of CEA expression are required (immunohistochemistry [IHC]2+ and IHC 3+). For CRC, pancreatic and gastric cancer participants, the CEA assessment will be performed retrospectively and the result is not needed to enroll the participant

Exclusion Criteria:

* Participants with a history or clinical evidence of central nervous system primary tumors or metastases including leptomeningeal metastases unless they have been previously treated, are asymptomatic, and have had no requirement for steroids or enzyme-inducing anticonvulsants in the last 14 days before screening
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for at least 2 weeks prior to enrollment
* Leptomeningeal disease
* Participants with paraspinal, paratracheal and mediastinal pathologic lesions larger than 2 centimeters unless they are previously irradiated. Irradiation of lesions must be completed at least 14 days prior to initiation of study treatment
* Participants with another invasive malignancy in the last 2 years (with the exception of basal cell carcinoma and tumors deemed by the investigator to be of low likelihood for recurrence)
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results or contraindicate the use of an investigational drug, including diabetes mellitus, history of relevant cardio-pulmonary disorders, and known autoimmune diseases
* Participants with bilateral lung lesions and dyspnea and/or with bilateral lung lesions and an oxygen saturation (SaO2) level less than 92% or participants with lobectomy or pneumonectomy with lung metastases in the remaining lung and either dyspnea or SaO2 less than 92% at baseline
* Uncontrolled hypertension (systolic blood pressure [BP] greater than [>] 150 millimeters of mercury [mmHg] and/or diastolic BP > 100 mmHg), unstable angina, congestive heart failure of any New York Heart Association classification, serious cardiac arrhythmia that requires treatment with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia, and history of myocardial infarction within 6 months of enrollment
* Active or uncontrolled infections
* Known human immunodeficiency virus (HIV) or known active hepatitis B or hepatitis C infection for participants not receiving obinutuzumab pretreatment
* Known HIV (HIV testing will be performed at screening if required by local regulations) in participants to be pretreated with obinutuzumab
* Pregnant or breastfeeding women
* Known hypersensitivity to any of the components of RO6958688 and/or obinutuzumab
* Concurrent therapy with any other investigational drug
* Last dose of any chemotherapy less than 28 days prior to the first RO6958688 infusion
* Expected need for regular immunosuppressive therapy
* Regular dose of corticosteroids the 28 days prior to Day 1 of this study or anticipated need for corticosteroids that exceeds prednisone 10 mg/day or equivalent within 28 days prior to the first RO6958688 infusion. Inhaled and topical steroids are permitted
* Radiotherapy within the last 28 days prior to the first RO6958688 infusion with the exception of limited-field palliative radiotherapy.

Additional Exclusion Criteria for Participants to be Pretreated with Obinutuzumab:

* Positive test results for human T-lymphotropic virus 1 (HTLV-1) or active HIV infection
* Positive test results for chronic hepatitis B infection or hepatitis C
* Known active tuberculosis (TB) requiring treatment within 3 years prior to baseline or latent TB that has not been appropriately treated
* Active bacterial, viral, fungal, or other infection, or any major episode of infection requiring treatment with intravenous (IV) antibiotics within 4 weeks of Cycle 1, Day 1
* Known hypersensitivity to any of the components of obinutuzumab; hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* History of progressive multifocal leukoencephalopathy (PML)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2019-09-03 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) or Serious Adverse Events (SAEs) | Baseline up to 60 months
Percentage of Participants with Dose-Limiting Toxicities (DLTs) | Day 1 up to Day 21
Percentage of Participants With Anti-Drug Antibodies (ADAs) Against RO6958688 | Pre-dose (Hour 0) on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome description section)
  Part I: Pre-dose (Hour 0) on Day 1 of Cycles 1, 2-3; 120 hours after end of infusion (EOI) in Cycle 1. Part II QW: pre-dose (Hour 0) on Day 1 of Cycles 1, 2, 3, 4. Part II Q3W: pre-dose (Hour 0) on Day 1 of Cycles 1, 2, 3, 4; 120 hours and 336 hours after EOI in Cycle 1, and 120 hours after EOI in Cycles 2, 3, 4. For Part I and II (QW and Q3W): pre-dose (Hour 0) on Day 1 of every cycle after Cycle 4 (Cycle 3 for Part I) up to treatment discontinuation (approximately 60 months), 28 days after last dose (approximately 60 months) (Cycle = 7 days for Part I and II QW; 21 days for Part II Q3W) (infusion duration = 30 minutes for Part I and 120 minutes for Part II [QW and Q3W])
MTD of RO6958688 With/Without Obinutuzumab Pretreatment | Day 1 up to Day 21
Late Cycle MTD of RO6958688 Without Obinutuzumab Pretreatment for the Step up Dosing Regimen | Day 1 up to Day 7 of each cycle as long as the dose is escalated weekly in Part II QW (up to approximately 60 months; Cycle = 7 days)
  Late cycle MTD is defined as the highest dose with less than or equal to DLT having been observed for 6 evaluable participants. If more than 6 participants are evaluable for DLT, late cycle MTD is the highest dose where less than (<) 33% of participants have DLT.
Maximum Serum Concentration (Cmax) for RO6958688 | Pre-dose (Hour 0) on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome description section)
  Part I: Pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2-3; 24, 48, and 120 hours after EOI of Cycle 1. Part II QW: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24 and 120 hours after EOI of Cycles 1 and 2; 48 hours after EOI of Cycle 1. Part II Q3W: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24, 48, 120, and 336 hours after EOI of Cycle 1; 24 and 120 hours after EOI of Cycles 2, 3, and 4; 48 hours after EOI of Cycle 2. For Part I and II (QW and Q3W): pre-dose (Hour 0), EOI, 2 hours after EOI (only for Part I) on Day 1 of every cycle after Cycle 4 (Cycle 3 for Part I), 2 hours after EOI on Day 1 of Cycles 8 and 12 (only for Part II QW) up to treatment discontinuation (approximately 60 months), 28 days after last dose (approximately 60 months) (Cycle =7 days for Part I and II QW; 21 days for Part II Q3W) (infusion duration = 30 minutes for Part I and 120 minutes for Part II [QW and Q3W])
Area Under the Concentration-Time Curve (AUC) for RO6958688 | Pre-dose (Hour 0) on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome description section)
  Part I: Pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2-3; 24, 48, and 120 hours after EOI of Cycle 1. Part II QW: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24 and 120 hours after EOI of Cycles 1 and 2; 48 hours after EOI of Cycle 1. Part II Q3W: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24, 48, 120, and 336 hours after EOI of Cycle 1; 24 and 120 hours after EOI of Cycles 2, 3, and 4; 48 hours after EOI of Cycle 2. For Part I and II (QW and Q3W): pre-dose (Hour 0), EOI, 2 hours after EOI (only for Part I) on Day 1 of every cycle after Cycle 4 (Cycle 3 for Part I), 2 hours after EOI on Day 1 of Cycles 8 and 12 (only for Part II QW) up to treatment discontinuation (approximately 60 months), 28 days after last dose (approximately 60 months) (Cycle =7 days for Part I and II QW; 21 days for Part II Q3W) (infusion duration = 30 minutes for Part I and 120 minutes for Part II [QW and Q3W])
Half-Life (t1/2) of RO6958688 | Pre-dose (Hour 0) on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome description section)
  Part I: Pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2-3; 24, 48, and 120 hours after EOI of Cycle 1. Part II QW: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24 and 120 hours after EOI of Cycles 1 and 2; 48 hours after EOI of Cycle 1. Part II Q3W: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24, 48, 120, and 336 hours after EOI of Cycle 1; 24 and 120 hours after EOI of Cycles 2, 3, and 4; 48 hours after EOI of Cycle 2. For Part I and II (QW and Q3W): pre-dose (Hour 0), EOI, 2 hours after EOI (only for Part I) on Day 1 of every cycle after Cycle 4 (Cycle 3 for Part I), 2 hours after EOI on Day 1 of Cycles 8 and 12 (only for Part II QW) up to treatment discontinuation (approximately 60 months), 28 days after last dose (approximately 60 months) (Cycle =7 days for Part I and II QW; 21 days for Part II Q3W) (infusion duration = 30 minutes for Part I and 120 minutes for Part II [QW and Q3W])
Clearance (CL) of RO6958688 | Pre-dose (Hour 0) on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome description section)
  Part I: Pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2-3; 24, 48, and 120 hours after EOI of Cycle 1. Part II QW: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24 and 120 hours after EOI of Cycles 1 and 2; 48 hours after EOI of Cycle 1. Part II Q3W: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24, 48, 120, and 336 hours after EOI of Cycle 1; 24 and 120 hours after EOI of Cycles 2, 3, and 4; 48 hours after EOI of Cycle 2. For Part I and II (QW and Q3W): pre-dose (Hour 0), EOI, 2 hours after EOI (only for Part I) on Day 1 of every cycle after Cycle 4 (Cycle 3 for Part I), 2 hours after EOI on Day 1 of Cycles 8 and 12 (only for Part II QW) up to treatment discontinuation (approximately 60 months), 28 days after last dose (approximately 60 months) (Cycle =7 days for Part I and II QW; 21 days for Part II Q3W) (infusion duration = 30 minutes for Part I and 120 minutes for Part II [QW and Q3W])
Volume of Distribution at Steady State (Vss) of RO6958688 | Pre-dose (Hour 0) on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome description section)
  Part I: Pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2-3; 24, 48, and 120 hours after EOI of Cycle 1. Part II QW: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24 and 120 hours after EOI of Cycles 1 and 2; 48 hours after EOI of Cycle 1. Part II Q3W: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24, 48, 120, and 336 hours after EOI of Cycle 1; 24 and 120 hours after EOI of Cycles 2, 3, and 4; 48 hours after EOI of Cycle 2. For Part I and II (QW and Q3W): pre-dose (Hour 0), EOI, 2 hours after EOI (only for Part I) on Day 1 of every cycle after Cycle 4 (Cycle 3 for Part I), 2 hours after EOI on Day 1 of Cycles 8 and 12 (only for Part II QW) up to treatment discontinuation (approximately 60 months), 28 days after last dose (approximately 60 months) (Cycle =7 days for Part I and II QW; 21 days for Part II Q3W) (infusion duration = 30 minutes for Part I and 120 minutes for Part II [QW and Q3W])
Minimum Drug Concentration (Cmin) for RO6958688 | Pre-dose (Hour 0) on Cycle 1 Day 1 up to 60 months (detailed timeframe is provided in outcome description section)
  Part I: Pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2-3; 24, 48, and 120 hours after EOI of Cycle 1. Part II QW: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24 and 120 hours after EOI of Cycles 1 and 2; 48 hours after EOI of Cycle 1. Part II Q3W: pre-dose (Hour 0), EOI, 2 hours after EOI on Day 1 of Cycles 1, 2, 3, and 4; 24, 48, 120, and 336 hours after EOI of Cycle 1; 24 and 120 hours after EOI of Cycles 2, 3, and 4; 48 hours after EOI of Cycle 2. For Part I and II (QW and Q3W): pre-dose (Hour 0), EOI, 2 hours after EOI (only for Part I) on Day 1 of every cycle after Cycle 4 (Cycle 3 for Part I), 2 hours after EOI on Day 1 of Cycles 8 and 12 (only for Part II QW) up to treatment discontinuation (approximately 60 months), 28 days after last dose (approximately 60 months) (Cycle =7 days for Part I and II QW; 21 days for Part II Q3W) (infusion duration = 30 minutes for Part I and 120 minutes for Part II [QW and Q3W])
Cmax for Obinutuzumab | Screening (pre-obinutuzumab dose [Hour 0] and EOI on Day -13 or Days -13 and -12), pre-RO6958688 dose [Hour 0] on Day 1 of Cycles 1, 2, 4, 8, and 12 in Part II QW (Cycle = 7 days)
Cmin for Obinutuzumab | Screening (pre-obinutuzumab dose [Hour 0] and EOI on Day -13 or Days -13 and -12), pre-RO6958688 dose [Hour 0] on Day 1 of Cycles 1, 2, 4, 8, and 12 in Part II QW (Cycle = 7 days)

SECONDARY OUTCOMES:
Percentage of Participants With an Objective Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1 | Baseline up to 60 months (detailed timeframe is provided in outcome description section)
  Baseline up to 60 months (assessed at Screening, at 12 weeks [in Part I], at 8 weeks [in Part II QW and Q3W] after Cycle 1 Day 1, every 8 weeks for the first 12 months, thereafter every 12 weeks until disease progression or death whichever occurs first, up to 60 months) (Cycle = 7 days for Part I and II QW, and 21 days for Part II Q3W)
Duration of Response (DOR) According to RECIST v1.1 | Baseline up to 60 months (detailed timeframe is provided in outcome description section)
  Baseline up to 60 months (assessed at Screening, at 12 weeks [in Part I], at 8 weeks [in Part II QW and Q3W] after Cycle 1 Day 1, every 8 weeks for the first 12 months, thereafter every 12 weeks until disease progression or death whichever occurs first, up to 60 months) (Cycle = 7 days for Part I and II QW, and 21 days for Part II Q3W)
Percentage of Participants With Stable Disease (SD) According to RECIST v1.1 | Baseline up to 60 months (detailed timeframe is provided in outcome description section)
  Baseline up to 60 months (assessed at Screening, at 12 weeks [in Part I], at 8 weeks [in Part II QW and Q3W] after Cycle 1 Day 1, every 8 weeks for the first 12 months, thereafter every 12 weeks until disease progression or death whichever occurs first, up to 60 months) (Cycle = 7 days for Part I and II QW, and 21 days for Part II Q3W)
Percentage of Participants With Disease Control, Defined as PR+CR+SD, According to RECIST v1.1 | Baseline up to 60 months (detailed timeframe is provided in outcome description section)
  Baseline up to 60 months (assessed at Screening, at 12 weeks [in Part I], at 8 weeks [in Part II QW and Q3W] after Cycle 1 Day 1, every 8 weeks for the first 12 months, thereafter every 12 weeks until disease progression or death whichever occurs first, up to 60 months) (Cycle = 7 days for Part I and II QW, and 21 days for Part II Q3W)
Progression-Free Survival (PFS) According to RECIST v1.1 | From the first study treatment to the first occurrence of objective disease progression or death from any cause (up to 60 months)
Change From Baseline in Activated Intra-Tumoral Cells | Baseline, Day 1 of Cycles 2, 3, 4, or 7 in Part II QW and Q3W (Cycle = 7 days for Part II QW and 21 days for Part II Q3W)
Best Overall Response (BOR) | Baseline up to 60 months (detailed timeframe is provided in outcome description section)
  Baseline up to 60 months (assessed at Screening, at 12 weeks [in Part I], at 8 weeks [in Part II QW and Q3W] after Cycle 1 Day 1, every 8 weeks for the first 12 months, thereafter every 12 weeks until disease progression or death whichever occurs first, up to 60 months) (Cycle = 7 days for Part I and II QW, and 21 days for Part II Q3W)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- United States (9):
  - Cedars Sinai Medical Center; Samuel-Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Stanford University, Palo Alto, California
  - UCLA Cancer Center, Santa Monica, California
  - University Of Colorado, Aurora, Colorado
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Dana Farber - Harvard, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - Sarah Cannon Cancer Center, Germantown, Tennessee
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Centre Leon Berard; Departement Oncologie Medicale, Lyon, France
- Italy (2):
  - IRCCS IST. Tumori Fondaz. Pascale; S.C. Oncologia Medica,Melanoma,Immunoterapia E Terapie Innovative, Napoli, Campania
  - Azienda Ospedaliera Universitaria Senese, U.O.C. Immunoterapia Oncologica, Siena, Tuscany
- Antoni van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- Spain (6):
  - Clinica Universitaria de Navarra; Servicio de Oncologia, Pamplona, Navarre
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - START Madrid-FJD, Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid

REFERENCES:
- [Derived] Martinez-Sabadell A, Morancho B, Rius Ruiz I, Roman Alonso M, Ovejero Romero P, Escorihuela M, Chicote I, Palmer HG, Nonell L, Alemany-Chavarria M, Klein C, Bacac M, Arribas J, Arenas EJ. The target antigen determines the mechanism of acquired resistance to T cell-based therapies. Cell Rep. 2022 Oct 18;41(3):111430. doi: 10.1016/j.celrep.2022.111430. PMID 36261015